CLINICAL TRIAL: NCT03425669
Title: Acoustic and Vestibular Noise as Possible Non-pharmacological Treatments of ADHD in School Children
Brief Title: Acoustic and Vestibular Noise as Possible Non-pharmacological Treatment of ADHD in School Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Sponsor
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: ADHD
Keywords: Acoustic and vestibular noise stimulation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: Patients will be recruited from Child and Adolescent Psychiatry in Lund and Malmö. Typically developing children (TDC) and inattentive children without diagnosis will be recruited from schools.
  All participants will perform a double-blind placebo cross over control study. ADHD participants will perform the entire test battery at three occasions with 2-3 weeks intermission in between tests. One occasion with placebo medication and sham SVS stimulation; one occasion with active SVS stimulation; and one occasion with active medication. TD children will only be tested twice and just perform under SVS vs. sham conditions.
  Test battery: 1) Episodic memory will be tested trough Auditory Verbal Learning Test (AVLT) (e.g. Dige et al., 2008). 2) Visuo-spatial working memory will be tested through the Spanboard task (Westerberg et al., 2004). 3) Motor-neurological investigation. 4) A finger tapping task. 5) Evaluation of an iPhone auditory noise application in a normal school setting.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be randomized to placebo or stimulant medication during assessments. Participants will be unaware if they will get sham stimulation or SVS (but not the test administrator).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo medication and sham stimulation (Active Comparator): Patients will be randomly chosen to the group who will get a combination of placebo and sham stimulation.
  Interventions: Device: Sham stimulation
- Active medication (Active Comparator): Patients are randomly chosen to the group who will get active medication without stimulation.
  Interventions: Drug: Active medication
- Active stimulation (Sham Comparator): Patients are randomly chosen to the group who will get acitive stimulation without taking medicine.
  Interventions: Device: Stochastic Vestibular Stimulation
- Controls with sham stimulation (Active Comparator): Controls without ADHD are randomly chosen to the group who will get sham stimulation.
  Interventions: Device: Sham stimulation
- Controls with active stimulation (Sham Comparator): Controls without ADHD are randomly chosen to the group who will get active stimulation.
  Interventions: Device: Stochastic Vestibular Stimulation

INTERVENTIONS:
Device: Stochastic Vestibular Stimulation — Stochastic vestibular stimulation will be given by electric stimulation through electrodes place over the mastoid processes behind each ear. Auditory stimulation with stochastic white noise will be administrated through ear phones.
  Other Names: Auditory white noise stimulation
  Arms: Active stimulation; Controls with active stimulation
Device: Sham stimulation — Patients will receive sham stimulation in place of active vestibular stimulation.
  Arms: Controls with sham stimulation; Placebo medication and sham stimulation
Drug: Active medication — Patients will be examined with and without medication.
  Other Names: Concerta, Ritalin, Methylphenidate, Equasym or Medikinet
  Arms: Active medication

SUMMARY:
Noise benefit in ADHD Auditory noise benefit: The original findings from our research group, that auditory noise enhances cognitive performance in inattentive children without diagnosis as well as children with an ADHD diagnosis, have been replicated several times (Baijot et al., 2016; Söderlund et al., 2016; Söderlund & Nilsson Jobs, 2016; Söderlund et al., 2007). In a new study, the benefit of noise was shown to be in parity with or even larger than the benefit of pharmacological ADHD treatment on two cognitive tasks, episodic word recall and visuo-spatial working memory task. In the study a group of children diagnosed with ADHD were tested on and off medication, at separate occasions, in noisy vs. silent environments while performing the tasks (Söderlund, Björk et al., 2016).

Participants and recruitment: Participants with an ADHD diagnosis using medication will be recruited from Child and Adolescent Psychiatry in Lund and Malmö. Typically developing children (TDC) and inattentive children without diagnosis will be recruited from schools in collaboration with the municipality.

Experimental design: All participants will perform a double-blind placebo cross over control study. ADHD participants will perform the entire test battery at three occasions with 2-3 weeks intermission in between tests. One occasion with placebo medication and sham SVS stimulation; one occasion with active SVS stimulation; and one occasion with active medication. TD children will only be tested twice while they will not be given any medication or placebo and just perform under SVS vs. sham conditions.

Test battery: 1) Episodic memory will be tested trough Auditory Verbal Learning Test (AVLT) (e.g. Dige et al., 2008). 2) Visuo-spatial working memory will be tested through the Spanboard task (Westerberg et al., 2004). 3) Motor-neurological investigation. 4) A finger tapping task. 5) Evaluation of an iPhone auditory noise application in a normal school setting. Our research group has developed an iPhone application (www.smartnoise.se) that is available at App-store right now. The study will last for about 5 months and participants will be 50 voluntary secondary school pupils that have documented attention difficulties as judged by their teachers. The application will be evaluated both by pupils, teachers and parents.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity disorder (ADHD) is one of the most frequent childhood disorders with an estimated prevalence of about 5-7% (e.g. Ullebo et al., 2012). Today the most common treatment approach is stimulant medication, e.g. methylphenidate (Greenhill et al., 2002; Wigal et al., 2011). However there are many concerns about medication: i) best dose for cognitive functioning and adapted school behavior differs (Hale et al., 2011), ii) it is not even evident that medication improves learning processes (Molina et al., 2009), iii) concerns regarding potential for drug abuse (Gordon et al., 2004); and iv) uncertainties regarding long term effects of drug use on the developing brain (Andersen, 2005).

In both national and international guidelines of ADHD care multimodal treatment is recommended (Young & Amarasinghe, 2010), but most patients only receive pharmacological treatment, sometimes in combination with parent training. If auditory or vestibular noise, as the present project suggests, could be a complement or an alternative to stimulant medication it could fundamentally change the treatment of ADHD and the school situation for those children.

Noise benefit in ADHD Auditory noise benefit: The original findings from our research group, that auditory noise enhances cognitive performance in inattentive children without diagnosis as well as children with an ADHD diagnosis, have been replicated several times (Baijot et al., 2016; Söderlund et al., 2016; Söderlund & Nilsson Jobs, 2016; Söderlund et al., 2007). In a new study, the benefit of noise was shown to be in parity with or even larger than the benefit of pharmacological ADHD treatment on two cognitive tasks, episodic word recall and visuo-spatial working memory task. In the study a group of children diagnosed with ADHD were tested on and off medication, at separate occasions, in noisy vs. silent environments while performing the tasks (Söderlund, Björk et al., 2016). Inattentive and low achieving school children have been shown to improve their memory recall when exposed to noise, whereas attentive and high achieving children perform worse during noise exposure (Helps et al., 2014; Söderlund & Sikström, 2008, 2012; Söderlund et al., 2010).

Vestibular noise benefit: Vestibular stimulation has since long been demonstrated to increase hippocampal activity and hippocampus is well demonstrated to be of crucial importance in detecting and holding on to spatial targets showing that hippocampus is of fundamental for both spatial orientation and learning in general (Moser et al., 2015). Therefore it is not surprising that external stochastic vestibular stimulation (SVS) exerts beneficial effects in different domains, e.g. balance in healthy astronauts (Mulavara et al., 2011), in Parkinson patients (Pal et al., 2009; Samoudi et al., 2014) and response times in continuous performance task (Yamamoto et al., 2005). The theory about noise benefit is thoroughly described by Sikström and Söderlund (2007). 1. The first objective is to systematically evaluate the effects of stochastic vestibular noise on cognitive task performance and to compare these results with the ones of stimulant medication using a double blind RCT (Random Control Trial) design.

The second objective is to implement a practical application, to evaluate if auditory noise can be beneficial in an every day school setting by the use of an iPhone application (see: www.smartnoise.se).

Participants and recruitment: Participants with an ADHD diagnosis using medication will be recruited from Child and Adolescent Psychiatry in Lund and Malmö. Typically developing children (TDC) and inattentive children without diagnosis will be recruited from schools in collaboration with the municipality.

Experimental design: All participants will perform a double-blind placebo cross over control study. ADHD participants will perform the entire test battery at three occasions with 2-3 weeks intermission in between tests. One occasion with placebo medication and sham SVS stimulation; one occasion with active SVS stimulation; and one occasion with active medication. TD children will only be tested twice while they will not be given any medication or placebo and just perform under SVS vs. sham conditions.

Test battery: 1) Episodic memory will be tested trough Auditory Verbal Learning Test (AVLT) (e.g. Dige et al., 2008). 2) Visuo-spatial working memory will be tested through the Spanboard task (Westerberg et al., 2004). 3) Motor-neurological investigation. 4) A finger tapping task. 5) Evaluation of an iPhone auditory noise application in a normal school setting. Our research group has developed an iPhone application (www.smartnoise.se) that is available at App-store right now. The study will last for about 5 months and participants will be 50 voluntary secondary school pupils that have documented attention difficulties as judged by their teachers. The application will be evaluated both by pupils, teachers and parents.

ELIGIBILITY:
Inclusion Criteria: Children and adolescents with a diagnosis of ADHD and control children without at diagnosis.

-

Exclusion Criteria: Intellectual disability, psychosis, severe depression or anxiety

-

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Spanboard task | Ten weeks
  Test of visuo-spatial working memory
AVLT | Ten weeks
  Auditory Verbal Learning Test
Go No- go test | Ten weeks
  Test of impulse inhibition

SECONDARY OUTCOMES:
Soft- signs test | Ten weeks
  Test of minor neurological deficits
Flower trail | Ten weeks
  Test of perception, fine motor function and motor planning
Finger tapping task | Ten weeks
  Test of timing

CONTACTS AND LOCATIONS:
Overall Officials: Peik Gustafsson, MD, PhD, Principal Investigator — Department of clinical sciences, Lund Uniersity
Locations (1):
- Child and Adolescent Psychiatry, Department of Clinical Sciences Lund, Lund University, Lund, Skåne County, Sweden